CLINICAL TRIAL: NCT00504218
Title: Detection and Treatment of Endocrine Abnormalities in Childhood Cancer Survivors and Hematopoitic Stem Cell Transplant Recipients
Brief Title: Detection and Treatment of Endocrine Abnormalities in Childhood Cancer Survivors and Hematopoietic Stem Cell Transplant Recipients
Status: Terminated | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070192; 07-CH-0192
Record Dates: First submitted 2007-07-18; First posted 2007-07-19 (Estimated); Last update posted 2018-12-03 (Actual); Status verified 2018-06-12

CONDITIONS: Hypopituitarism; Hypogonadism; Thyroid Dysfunction; Bone Diseases, Metabolic
Keywords: Growth Factor; Hypothalamic-Pituitary Dysfunction; Primary Disorders of the Thyroid; Decreased Bone Mineral Density; Endocrine Side Effects Related to Cancer Therapy; Primary Gonadal Dysfunction; Obesity; Impaired Glucose Tolerance; Thyroid Disorder; Cancer Therapy Endocrine Side Effects; Pituitary Dysfunction; Childhood Cancer Survivors
MeSH Terms: conditions — Hypopituitarism; Hypogonadism; Bone Diseases, Metabolic; Obesity; Glucose Intolerance; Thyroid Diseases

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
This study will determine the prevalence of endocrine-related side effects in children who have been treated for cancer and establish a database and registry organized according to cancer diagnosis, treatments and endocrine side effects. In children, the endocrine system, which includes glands and hormones that help to control metabolism, growth, development and reproduction, is particularly vulnerable to long-term side effects associated with cancer and its treatments. The study will also serve to help train medical fellows, residents and students in identifying and managing endocrine abnormalities in children who have been diagnosed with and treated for cancer.

Children between 2 and 24 years of age who have been treated for a childhood cancer and have been disease-free for at least 1 year may be eligible for this study.

All participants undergo the following procedures:

* Review of cancer treatment record
* Review of medical and family history
* Blood draw for DNA studies
* Physical examination and body measurements (height, weight, waist, body proportions)
* Completion of child health questionnaires
* Individualized screening and counseling program
* Review of the following endocrine systems: growth, pituitary and hypothalamic function, thyroid function, ovary and testicular function, bone health, risk of obesity and diabetes

The following additional studies may be done, as clinically indicated:

* Magnetic resonance imaging (MRI) of the brain
* Thyroid, testicular or ovarian ultrasound
* DEXA scan to measure bone density
* Wrist x-ray to measure bone age
* Blood tests
* Urine pregnancy test for girls who are old enough to have menstrual periods
* Stimulation testing (tests that involve giving medicine by mouth or in the vein and then measuring blood levels of substances afterwards, such as oral glucose tolerance test, arginine-clonidine growth hormone stimulation test, ACTH stimulation test, and gonadotropin-releasing hormone stimulation test)

Children with endocrine abnormalities are offered standard treatments.

DETAILED DESCRIPTION:
Endocrine dysfunction is increasingly recognized as one of the most important aspects of quality of life issues, physical and psychosocial development and overall prognosis in pediatric patients diagnosed with neoplasms as well as in patients s/p bone marrow transplant throughout their lifespan. In addition, several of the new, molecularly designed therapies for neoplasms may interact with endocrine signaling; these include receptors and/or their ligands for growth and/or proliferation factors, and disruptors of steroid hormone interactions. The present study serves as a natural history protocol.

As a natural history, this protocol allows our Institute to care for pediatric and adult patients with endocrine related complications associated with prior cancer therapy and/or hematopoietic stem cell transplant (HSCT) for the purposes of:

Training our fellows, residents and students in the identification and management of endocrine abnormalities developing in patients who have been diagnosed with and treated for neoplasms and/or who have received HSCT at the NIH-Clinical center.

Developing new clinical studies for the recognition and therapy of endocrine side effects related to cancer therapy and/or HSCT: this protocol will eventually lead to new, separate protocols that will address specific aspects of endocrinopathies in childhood cancer survivors and HSCT survivors.

The protocol will serve as the basis for outpatient clinics that will function within the context of the pediatric and adult endocrine outpatient clinics: every eligible patient referred to the endocrine service from the NCI, NHLBI, and other NIH institutions and centers will be enrolled in this study, which for the first time will create an endocrine database for these patients. As stated in our aims above, it is our hope that the present investigation will serve as an incubator of further research-focused studies with the ultimate goal of improving the life of children and adults who have been cured of their underlying neoplasms as well as those individuals who are recipients of an HSCT.

ELIGIBILITY:
* INCLUSION
* Age >2 years.
* History of diagnosis of malignancy or HSCT and completion of therapy prior to entering the study. Eligible patients must be free of their underlying malignancy for at least one year prior to entering the study, as confirmed by records from the referring oncologist.
* We will request permission to administer the Child Health Questionnaires (PF 50 and CF87) to all patients who are enrolled in this protocol. This instrument has been validated for use in children ages five and older. Children 10 years and older will complete the child version. The Child Health Questionnaire (CHQ) has been normed in a representative sample in the US, and is being used in large population studies in Australia, Ireland, and the UK. Additionally, it has been rigorously translated into a number of languages using international guidelines including American-Spanish, Canadian-French, Dutch, Finnish, French, German, Italian, Greek, Honduran-Spanish, Mexican-Spanish, Norwegian, Portuguese, and Swedish. For this study will purchase the CHQ in American- Spanish in order to include Spanish-speaking subjects in this part of the study. The costs to purchase the CHQ in numerous languages would be prohibitive for this pilot study. However, if a significant number of subjects in a specific language are recruited, we will consider the purchase of the CHQ for that group of subjects.

EXCLUSION FOR CAROTID MRI

* Metal implants or other ferromagnetic devices, or Foreign material
* Claustrophobia

Ages: 2 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2007-07-17; Study Completion 2018-06-12

CONTACTS AND LOCATIONS:
Overall Officials: Maya B Lodish, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Jemal A, Murray T, Samuels A, Ghafoor A, Ward E, Thun MJ. Cancer statistics, 2003. CA Cancer J Clin. 2003 Jan-Feb;53(1):5-26. doi: 10.3322/canjclin.53.1.5. PMID 12568441
- [Background] Oeffinger KC, Mertens AC, Sklar CA, Kawashima T, Hudson MM, Meadows AT, Friedman DL, Marina N, Hobbie W, Kadan-Lottick NS, Schwartz CL, Leisenring W, Robison LL; Childhood Cancer Survivor Study. Chronic health conditions in adult survivors of childhood cancer. N Engl J Med. 2006 Oct 12;355(15):1572-82. doi: 10.1056/NEJMsa060185. PMID 17035650
- [Background] Cohen LE. Endocrine late effects of cancer treatment. Endocrinol Metab Clin North Am. 2005 Sep;34(3):769-89, xi. doi: 10.1016/j.ecl.2005.04.008. PMID 16085170